CLINICAL TRIAL: NCT06388070
Title: A Multicenter, Randomized, Double-blinded, Non-inferiority Phase 3 Study to Evaluate the Efficacy and Safety of HUC3-053 Compared With Hyalein Mini Eye Drops in Patients With Dry Eye Syndrome
Brief Title: To Evaluate the Efficacy and Safety of HUC3-053 in Patients With Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUC3-053
Record Dates: First submitted 2024-04-10; First posted 2024-04-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HUC3-053 (Experimental): Participants received "HUC3-053" drops in each eye five to six times a day for 12 weeks.
  Interventions: Drug: HUC3-053
- Hyalein Mini Drops (Active Comparator): Participants received "Hyalein Mini Drops" in each eye five to six times a day for 12 weeks.
  Interventions: Drug: Hyalein Mini Drops

INTERVENTIONS:
Drug: HUC3-053 — drops in each eye five to six times a day for 12 weeks
  Other Names: Kynex 3 eye drops
  Arms: HUC3-053
Drug: Hyalein Mini Drops — drops in each eye five to six times a day for 12 weeks.
  Other Names: Hyalein Mini Drops 0.3%
  Arms: Hyalein Mini Drops

SUMMARY:
This is a multi-center, randomized, double-blinded, non-inferiority study to evaluate the efficacy and safety of HUC3-053 in patients with dry eye syndrome.

After a 2-week run-in period, patients will be randomized equally to the HUC3-053 or Hyalein Mini Drops administered bilaterally five to six times a day for 12 weeks.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blinded, non-inferiority study to evaluate the efficacy and safety of HUC3-053 in patients with dry eye syndrome.

During a 2-week study run-in period prior to randomization, all subjects will receive rescue drug bilaterally up to 4 times a day. Randomization will then occur as 1:1 where patients will be assigned to receive HUC3-053 or Hyalein Mini Drops given bilaterally five to six times a day. The treatment period is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age over 19
* Volunteer who have had more than one symptom of dry eye disease for at least 3 month before screening visit.
* Corneal staining score(Oxford grading) ≥ 2 and Schirmer test ≤ 10mm/5min (If Schirmer test = 0mm/5min, Nasal stimulation schirmer test ≥ 3mm/5min) and TBUT test ≤10 and OSDI (Ocular Surface Disease Index) ≥ 23 in at least one of both eyes
* Best corrected visual acuity ≥ 0.2 in both eyes at Screening and Randomization Visit

Exclusion Criteria:

* The patients with clinically significant ocular disorders affected the test result Current or recent patients used dry eye syndrome medications (topical or systemic) that may affect the status
* SBP ≥140mmHg or DBP ≥ 90mmHg or HbA1c>9%
* Wearing contact lenses within 72 hr of screening visit
* Pregnancy or Breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Corneal staining score | Week 12
  Change from Baseline in Corneal staining score at week 12

SECONDARY OUTCOMES:
Change from Baseline in Corneal staining score | Week 4, 8
  Change from Baseline in Corneal staining score at week 4, 8
Change from Baseline in Conjunctival staining score | Week 4, 8, 12
  Change from Baseline in Conjunctival staining score at week 4, 8, 12
Change from Baseline in Schirmer test | Week 4, 8, 12
  Change from Baseline in Schirmer test at week 4, 8, 12
Change from Baseline in Tear film break-up time | Week 4, 8, 12
  Change from Baseline in Tear film break-up time at week 4, 8, 12
Change from Baseline in Ocular surface disease index | Week 4, 8, 12
  Change from Baseline in Ocular surface disease index at week 4, 8, 12
Change from Baseline in Eye Soreness after eye drop assessed by NRS | Week 4, 8, 12
  Change from Baseline in Eye Soreness after eye drop assessed by NRS at week 4, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Chul Young Choi, Principal Investigator — Gangbuk Samsung Hospital
Locations (1):
- Gangbuk Samsung Hospital, Seoul, Jongno-gu, South Korea